CLINICAL TRIAL: NCT02517138
Title: Right-front Direction in Parabolic Flight
Acronym: DROITDEVANT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 11-094
Record Dates: First submitted 2015-07-23; First posted 2015-08-06 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Healthy
Keywords: volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Measurements of eye movements and perception (Other)
  Interventions: Other: Parabolic flight; Other: Measurements of eye movements and perception

INTERVENTIONS:
Other: Parabolic flight
Other: Measurements of eye movements and perception

SUMMARY:
The goal of this study is to objectively determine the perceived direction of the right-front by the subjects in weightlessness. The direction of the right-front has not been investigated to date with the measurements of the position of the eyes. The investigators will compare the intersection of the horizontal and vertical saccadic trajectories (jerky) with the apparent direction of the right-front indicated by the subjects when they look right front in the dark (LOOK) and that they indicate when they determine whether a visual target through the right-front apparent (PERCEPTION). Then, the investigators will compare these measurements between normal gravity and microgravity hypergravity during parabolic flight.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (men or women)
* Aged between 20-65 years
* Affiliates to a social security system
* Who are willing to take part in the study,
* Who gave written informed consent,
* Declared fit after a similar visit to a medical aeronautical medical fitness for the non-professional cabin crew in civil aviation. There will be no other aptitude tests for the selection of subjects.

Exclusion Criteria:

* People who participated in a biomedical research protocol for which the exclusion period is complete,
* pregnant women.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-11; Primary Completion 2013-03 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
eye movements | Baseline
  measurements between normal gravity and microgravity hypergravity during parabolic flight
acceleration of the head | Baseline
  measurements between normal gravity and microgravity hypergravity during parabolic flight
perception by the subjects of the right-front. | Baseline
  measurements between normal gravity and microgravity hypergravity during parabolic flight
acceleration of the arms | Baseline
  measurements between normal gravity and microgravity hypergravity during parabolic flight

CONTACTS AND LOCATIONS:
Locations (1):
- Umr Ucbn/Inserm U1075 Comete, Caen, Basse-Normandie, France